CLINICAL TRIAL: NCT04696861
Title: Telehealth to Reduce Suicidality and Improve HIV Care Engagement in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00107424; K08MH124459 (NIH)
Record Dates: First submitted 2020-12-22; First posted 2021-01-06 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-09

CONDITIONS: Suicide; Suicidal Ideation; HIV Infections; Adherence, Medication; Treatment Adherence and Compliance; Stigma, Social; Disclosure; Quality of Life
MeSH Terms: conditions — Suicide; Suicidal Ideation; HIV Infections; Medication Adherence; Treatment Adherence and Compliance; Social Stigma

STUDY DESIGN:
Intervention Model Description: Patients who screen positive for suicidal ideation will be enrolled in the study, complete the baseline survey, and then randomly assigned to the intervention (3 sessions of counseling) or enhanced standard of care (brief safety planning).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IDEAS for Hope Intervention (Experimental): Participants will receive three counseling sessions at two week intervals, delivered by telehealth by a trained psychiatric nurse, focused on managing suicidal ideation and enhancing HIV care engagement.
  Interventions: Behavioral: IDEAS for Hope
- Enhanced Standard of Care with Safety Planning (Active Comparator): Participants will receive a brief, 10-15 minute counseling session, delivered by telehealth by a trained psychiatric nurse, focused on safety planning.
  Interventions: Behavioral: Enhanced Standard of Care (Safety Planning)

INTERVENTIONS:
Behavioral: IDEAS for Hope — Participants will receive three counseling sessions at two week intervals, delivered by telehealth by a trained psychiatric nurse, focused on managing suicidal ideation and enhancing HIV care engagement.
  Arms: IDEAS for Hope Intervention
Behavioral: Enhanced Standard of Care (Safety Planning) — Participants will receive a brief, 10-15 minute counseling session, delivered by telehealth by a trained psychiatric nurse, focused on safety planning.
  Arms: Enhanced Standard of Care with Safety Planning

SUMMARY:
The overall objectives of the proposed research are to develop a brief telehealth counseling intervention to provide support for people living with HIV and experiencing suicidal ideation, and to support HIV care engagement. The investigators hypothesize that a brief telehealth counseling intervention will be safe (participants in the clinical trial will not have increased risk of suicidal behavior), acceptable (high patient retention and satisfaction, high fidelity), and will demonstrate preliminary efficacy (reduced suicidal ideation, improved care engagement, improved mental well-being).

DETAILED DESCRIPTION:
The objective of the proposed research is to assess the feasibility and acceptability of a 3-session, nurse-delivered telehealth intervention to reduce suicidality and improve HIV care engagement among adults living with HIV in the Kilimanjaro Region of Tanzania. Suicide is a leading cause of death among people living with HIV (PLWH) worldwide and mental health disorders are key contributors to poor HIV care engagement, lower quality of life, higher transmission risk, and increased mortality among PLWH. Conversely, connecting PLWH with targeted mental health support improves these critical health outcomes. Telehealth counseling represents a cost-effective, innovative approach to mental health treatment in low-resource settings such as Tanzania, with the potential to expediently extend services. The proposed study will include Aim 1: Identifying the desired characteristics of a telehealth intervention for suicidality and HIV care engagement in the Tanzanian clinical context, Aim 2: Refining intervention content with support from a local study advisory board in Tanzania, and Aim 3: Testing the telehealth model in a pilot randomized control trial. Given emerging evidence for telehealth approaches to improve access to treatment and reduce health disparities, the intervention has great potential to support NIMH strategic objectives to address mental health comorbidities and strengthen the HIV care continuum.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Attending HIV care at study clinic
* Screen positive for suicidal ideation
* Able to understand Kiswahili or English
* Medically stable
* Capable of providing informed consent to participate

Exclusion Criteria:

* Under 18 years old
* Unable to understand Kiswahili or English
* Experiencing medical or psychiatric symptoms requiring immediate treatment
* Incapable of providing informed consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Tanzania (2):
  - Majengo Health Centre, Moshi
  - Mawenzi Hospital, Moshi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madundo K, Mwobobia JM, Perry M, Knippler E, Amiri I, Msoka EF, Tarimo CS, Katiti V, Mmbaga BT, Goldston DB, Relf MV, Knettel BA. HIV and mental health provider experiences of implementing brief depression and suicide screening among people living with HIV in Tanzania: A qualitative study. PLOS Ment Health. 2025 Mar 13;2(3):e0000268. doi: 10.1371/journal.pmen.0000268. eCollection 2025. PMID 41661889
- [Derived] Knettel BA, Madundo K, Amiri I, Msoka EF, Pan W, Khofi T, Ngangula P, Turner EL, Joel L, Rwakilomba J, Tarimo CS, Katiti V, Knippler ET, Mmbaga BT, Relf MV, Goldston DB. Results of a Pilot Randomized Controlled Trial of IDEAS for Hope: A Brief Telehealth Intervention for Suicide Prevention and HIV Care Engagement in Tanzania. J Acquir Immune Defic Syndr. 2025 Dec 15;100(5):435-444. doi: 10.1097/QAI.0000000000003758. PMID 40905305

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Started | 30 | 30
Completed | 26 | 30
Not Completed | 4 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.83 (11.86) | 42.67 (10.99) | 43.25 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 30 | 60
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Suicidal Ideation
Description: Columbia-Suicide Severity Rating Scale (C-SSRS) items measuring suicidal thoughts (yes/no), intent (yes/no), and plan (yes/no). Reported here are the number of participants who responded 'yes' to each of the items.
Time Frame: 3 months post enrollment
Population: 1 intervention participant died prior to 3-month follow-up and 1 intervention participant was lost to follow-up and did not complete the 3-month follow-up survey
Measure: Count of Participants; unit: Participants
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
Participants
  Suicidal Thoughts | 4 | 3
  Plan | 0 | 0
  Intent | 0 | 0
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; Generalized linear mixed models were conducted and odds ratios (ORs) were reported; Test type: Superiority; p = 0.961, Mixed Models Analysis — Unitized unadjusted bivariate analyses instead of adjusted multivariable analysis. This was a pilot study to estimate the magnitude of effect sizes for informing further large interventions. The significance level was also not adjusted

2. Primary Outcome: Number of Participants With a Gap in HIV Care Engagement
Description: Participant medical records were reviewed after the 3-month follow-up survey to identify whether they had a gap in care during the study period, defined as 6 or more days where they did not have enough prescribed medication on hand to maintain adherence between HIV clinic appointments.
Time Frame: 3 months post enrollment
Population: 1 intervention participant died prior to 3-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 29 | 30
Participants | 2 | 1
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; Generalized linear mixed models were conducted and odds ratios (ORs) were reported; Test type: Superiority; p = 0.961, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: HIV Medication Adherence, as Measured by Number of Participants Who Report Adherence Challenges
Description: During the baseline and follow-up surveys, participants were asked two questions related to their adherence to antiretroviral medication: "Think about the last 14 days. On how many days did you miss taking your HIV pill(s)?" and the same question with a 90 day recall period. Adherence challenges were coded yes/no at each time point, defined as (1) missing 3 or more days of medication in the past 14 days or (2) missing 6 or more days in the past 90 days.
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
Participants | 1 | 2
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; Generalized linear mixed models were conducted and odds ratios (ORs) were reported; Test type: Superiority; p = 0.368, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: Viral Load
Description: Extraction of routine HIV viral load testing from the patient medical record at baseline and 3-months post study enrollment.
Time Frame: Baseline, 3 months Post Enrollment
Population: Data not collected.
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Depression
Description: Patient Health Questionnaire (PHQ-9), 9 items, score 0-27 with higher indicating more depression
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 2.71 (2.43) | 3.13 (2.87)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; General linear mixed models; Test type: Superiority; p = 0.634, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: HIV Stigma
Description: HIV Stigma Scale (HSS), 12 items, score 12-48 with higher indicating more stigma
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 29.35 (3.49) | 30.31 (5.39)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; General linear mixed models; Test type: Superiority; p = 0.832, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of HIV Disclosures Made by Participants
Description: Self-reported disclosures to partner, family, friends, others (yes/no)
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Number; unit: Disclosures
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
Disclosures
  Disclosed to partner | 2 | 1
  Disclosed to family | 0 | 2
  Disclosed to friends | 4 | 2
  Disclosed to others | 0 | 2

8. Secondary Outcome: Total Number of HIV Disclosures Made by Participants
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Number; unit: Disclosures
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
Disclosures | 6 | 7
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; Generalized linear mixed models were conducted and odds ratios (ORs) were reported; Test type: Superiority; p = 0.624, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Social Support
Description: Perceived Availability of Support Scale (PASS), 7 items, score 7 to 35 with higher indicating more social support
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 27.21 (7.15) | 27.9 (7.42)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; General linear mixed models; Test type: Superiority; p = 0.833, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Acceptability of Intervention
Description: 10 items adapted from the Client Satisfaction Questionnaire (CSQ), score 10 to 40 with higher indicating greater satisfaction with the intervention
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 34.93 (3.11) | 33.5 (2.78)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; General linear mixed models; Test type: Superiority; p = 0.7, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Hopelessness
Description: Beck Hopelessness Scale (Balsamo Short Form), 9 items, score 0 to 9 with higher indicating more hopelessness
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 1.75 (2.12) | 2.4 (2.33)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; General linear mixed models; Test type: Superiority; p = 0.79, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

12. Secondary Outcome: Reasons for Living
Description: Brief Reasons for Living Inventory, 12 items, score 12 to 72 with higher indicating more reasons to live
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 60.54 (8.79) | 62.3 (5.49)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; General linear mixed models; Test type: Superiority; p = 0.55, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

13. Secondary Outcome: Quality of Life (Overall)
Description: The World Health Organization Quality of Life Brief Version (WHOQOL-BREF), 2 items, score 2 to 10 with higher indicating better quality of life
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 3.54 (0.84) | 3.60 (0.62)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; Test type: Superiority; p = .823, Mixed Models Analysis

14. Secondary Outcome: Quality of Life (Health Satisfaction)
Description: as for outcome 13
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 3.79 (0.74) | 3.73 (0.91)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; Test type: Superiority; p = .942, Mixed Models Analysis

15. Post Hoc Outcome: Anxiety
Description: Brief Symptom Inventory Anxiety Subscale, 6 items, score 0 to 24 with higher indicating more anxiety
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 5.5 (4.22) | 7.43 (5.71)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; General linear mixed models; Test type: Superiority; p = 0.207, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

16. Post Hoc Outcome: Suicide Coping Self-Efficacy
Description: Self-Efficacy to Avoid Suicidal Action (SEASA) Scale, 6 items, score 0 to 60 with higher indicating more coping self-efficacy
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 45.86 (11.51) | 43.53 (11.99)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; General linear mixed models; Test type: Superiority; p = 0.594, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

17. Post Hoc Outcome: Attitudes About Antiretroviral Therapy
Description: Beliefs About Medicine Questionnaire (BMQ), 10 items, score 10 to 50 with higher indicating more positive attitudes about medication
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 42.25 (3.53) | 42.73 (4.59)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; General linear mixed models; Test type: Superiority; p = 0.738, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

18. Post Hoc Outcome: HIV Acceptance
Description: Illness Cognition Questionnaire (ICQ), 7 items, score 7-28 with higher indicating more acceptance
Time Frame: 3 months post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
Number analyzed (Participants) | 28 | 30
score on a scale | 20.75 (2.77) | 20.73 (3.86)
Statistical Analysis 1: Comparison: IDEAS for Hope Intervention vs Enhanced Standard of Care With Safety Planning; General linear mixed models; Test type: Superiority; p = 0.845, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 3 months post enrollment
Description: One adverse event, a serious adverse event involving the death of a study participant, was reported to the study IRBs and determined to be not related to the study.
Arm/Group | IDEAS for Hope Intervention | Enhanced Standard of Care With Safety Planning
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDEAS for Hope Intervention (N=30) | Enhanced Standard of Care With Safety Planning (N=30)
AIDS-related complications (Immune system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT04696861/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT04696861/ICF_000.pdf